CLINICAL TRIAL: NCT03609970
Title: Vitamin D and Immunity: Photosynthesis Versus Supplementation
Acronym: IMMUNI-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RJ115/N204
Record Dates: First submitted 2018-06-22; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; UVR; Immune system
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- UVR (Solar simulated radiation) (Experimental): Twice weekly 1.25 SED (sub-erythemal) (4 weeks)
  Interventions: Radiation: UVR (Solar simulated radiation)
- Vitamin D3 supplementation (Experimental): 4X 1000IU cholecalciferol tablets daily (28 days)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Daily 4X 1000IU cholecalciferol
  Arms: Vitamin D3 supplementation
Radiation: UVR (Solar simulated radiation) — 1.25 SED Solar simulated radiation twice weekly
  Arms: UVR (Solar simulated radiation)

SUMMARY:
The optimal way to restore serum 25-hydroxyvitamin D sufficiency is currently debatable. UV irradiation through sunshine exposure promotes endogenous vitamin D synthesis, although this can also be associated with a risk of UVR-induced skin cancer. Dietary supplements represent an alternative, which are increasingly being used in clinical trials to correct deficiency. However, it is unclear whether sunshine exposure and vitamin D supplementation induce comparable changes in immune function, or whether additional UVR-induced molecules may be responsible for proposed health benefits. Several studies report an inverse correlation between exposure to UVR and immune-mediated diseases, further supporting the theory that UVR may also be protective through non vitamin-D mediated pathways. So far it has been difficult to distinguish between immune-regulation by vitamin D and other mediators induced by UVR as the downstream effects are similar. A direct comparison of the biological effects of vitamin D obtained by UVR versus supplementation has never been made. This study aims to elucidate the differences in vitamin D generated by UVR exposure versus supplementation by comparing immunological endpoints

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Fitzpatrick skin type I/II
* Healthy
* Serum 25(OH)D3 <50nmol/L

Exclusion Criteria:

Serum 25(OH)D3 >50nmol/L

* Pregnant or nursing women
* Women of child bearing age not using adequate contraception
* Are taking photosensitizing medication (i.e. causes you to be more sensitive to sunlight)
* Have had a history of skin disorders, sensitive skin, sensitivity to sunlight or skin cancer
* Have previously had an organ transplant
* Have partaken in a clinical study within the last 14 days
* Have had recent exposure to sunbeds (last 4 months) or holiday sun (including skiing)
* Are currently or have taken vitamin D supplements in the last 4 months Are asthmatic or suffer from any allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Vitamin D status of healthy participants treated with oral vitamin D (cholecalciferol) or UVR (SSR) exposures and control (untreated) | 3 years
  Measure 25(OH)D3nmol/L via LC-MS/MS

SECONDARY OUTCOMES:
Changes to peripheral blood cell frequency | 3 years
  Frequency of major peripheral immune cells (e.g. CD3+ T cells, CD3+ CD4+ T cells, CD3+ CD8+ T cells, CD19+ B cells, Natural Killer Cells, Classical, Non-classical and Intermediate Monocytes) in participants when vitamin D insufficient and sufficient. Via flow cytometry.
Impact upon the frequency and phenotype of peripheral blood dendritic cells | 3 years
  Frequency of peripheral blood dendritic cells (myeloid and plasmacytoid) in individuals with insufficient vitamin D levels and following vitamin D repletion via supplementation or UVR (SSR) exposures. Assessment of markers of maturation/tolerogenicity (MFI and frequency expressing) on myeloid and plasmacytoid dendritic cells direct ex vivo and after stimulation in vitro in participants when vitamin D insufficient and sufficient.
Gene expression in peripheral blood myeloid and plasmacytoid dendritic cells | 3 years
  Differentially regulated genes in myeloid and plasmacytoid dendritic cells in participants after vitamin D repletion via supplementation and UVR (SSR) exposure via Microarray.

CONTACTS AND LOCATIONS:
Overall Officials: Antony Young, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No